CLINICAL TRIAL: NCT05024916
Title: The Effect of Blueberry Consumption on Brain Health in Older Adults: in Vivo Measures of Cerebral Antioxidant and Cerebral Blood Flow
Brief Title: Blueberry Intervention Study for Brain Aging
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Kansas Medical Center (Other)
Collaborators: U.S. Highbush Blueberry Council (Other)
Responsible Party: Principal Investigator, In-Young Choi, Ph.D., Professor of Neurology, University of Kansas Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: STUDY00147614
Record Dates: First submitted 2021-08-23; First posted 2021-08-27 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-05

CONDITIONS: Brain Aging
MeSH Terms: interventions — Methods

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Experimental): Participants will receive the dietary intervention. Participants will take 1 serving of blueberries/day.
  Interventions: Dietary Supplement: Intervention
- Control (Active Comparator): Participants will receive a placebo. Participants will take 1 serving of placebo/day.
  Interventions: Dietary Supplement: Control

INTERVENTIONS:
Dietary Supplement: Intervention — 26 g packets of freeze-dried blueberries (equivalent to 1 cup of fresh blueberries) will be given to participants to be consumed daily. Participants will be asked to consume 1 packet per day for 3 months.
  Other Names: Freeze-dried blueberries
  Arms: Intervention
Dietary Supplement: Control — 26 g packets of isocaloric carbohydrate-matched powder will be given to participants to be consumed daily. Participants will be asked to consume 1 packet/day for 3 months.
  Other Names: Placebo
  Arms: Control

SUMMARY:
The purpose of this study is to determine if increased blueberry intake helps increase brain antioxidant (glutathione) and cerebral blood flow in older adults.

DETAILED DESCRIPTION:
Consuming blueberries may improve brain health of older adults by increasing the antioxidant levels in the brain to protect nerve cells in the aging brain. Researchers think that there may be a relationship between the brain's antioxidant defense system and blueberry intake due to the high antioxidant content in blueberries.

This study will investigate if blueberry intake may aid in enhancing glutathione levels and cerebral blood flow using special Magnetic Resonance Imaging (MRI) scans.

Participants will be asked to make a total of up to 4 visits to the research site. Participation will last about 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Speak English as the primary language and be able to read and write.
* Good general health with no concomitant diseases
* Low berry consumption (≤1 serving/week)
* Cognitively normal (Mini-Mental State Exam Score ≥24)
* BMI range=18.5-35 kg/m2.

Exclusion Criteria:

* Presence of any central neurological diseases or prior major head trauma with loss of consciousness
* Presence of an active unstable and life-threatening systemic illness
* Presence of major psychiatric disorders within the past 3 years including depression, anxiety, and alcohol or drug abuse
* Presence of diabetes mellitus; metabolic syndrome or uncontrolled hypertension
* Use of psychoactive and investigational medications
* MRI contraindications (pacemaker, aneurysm clips, artificial heart valves, metal fragments, foreign objects or claustrophobia)
* Blueberry or salicylate allergy
* Pregnancy

Ages: 65 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 63 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2024-10-03 (Actual); Study Completion 2024-10-03 (Actual)

PRIMARY OUTCOMES:
Change in brain glutathione (GSH) levels | Change from baseline to 3 months
  Measure of brain GSH with a 3 T MRI scanner
Change in cerebral blood flow (CBF) | Change from baseline to 3 months
  Measure of CBF with a 3 T MRI scanner

CONTACTS AND LOCATIONS:
Overall Officials: In-Young Choi, PhD, Principal Investigator — Department of Neurology
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States

IPD SHARING:
Plan to Share IPD: No